CLINICAL TRIAL: NCT05880498
Title: Smartphone Mindfulness Autism Research Team Study
Brief Title: Smartphone Mindfulness Autism Research Study
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2105000376
Record Dates: First submitted 2023-05-05; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Anxiety; Stress
Keywords: Autism; Mindfulness
MeSH Terms: conditions — Anxiety Disorders; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Intervention (Experimental): 6 week smartphone-based self-guided mindfulness training using a customized version of the Healthy Minds app.
  Participants were instructed to listen to at least one activity per day for 5 days per week, for 6 weeks. Activities that were part of the structured curriculum consisted of alternating mindfulness didactic 'lessons' (each up to 7 minutes in length) and mindfulness 'practices' (either 10 minutes or 15 minutes in length- as chosen by the participant).
  Interventions: Behavioral: Mindfulness Intervention
- Wait-List Control (WLC) (No Intervention): No intervention was administered during the 6-week wait list control period.

INTERVENTIONS:
Behavioral: Mindfulness Intervention — Self-guided mindfulness training using a customized version of the Healthy Minds app
  Arms: Mindfulness Intervention

SUMMARY:
Individuals diagnosed with autism are also often diagnosed with anxiety disorders. Therefore, having useful strategies to manage stress and anxiety may be particularly helpful for autistic individuals. Mindfulness-based interventions, delivered in-person as well as those offered remotely online, have been found to lower stress and anxiety. Although in-person mindfulness training has been found to be helpful for autistic individuals, there is little research that has studied remote app-based mindfulness training in autistic adults.

This study examines whether a six-week structured intervention, using a mindfulness app, lowers anxiety and stress in autistic adults. Participants were randomly assigned either to an intervention group, which started the intervention immediately, or a wait-list control group, which participated in the same intervention program six-weeks later. Findings will provide important information about the potential for remote app-based mindfulness training to lower stress and anxiety in adults diagnosed with autism.

DETAILED DESCRIPTION:
A significant proportion of individuals diagnosed with autism are also diagnosed with one or more anxiety disorders. Since stress and anxiety in autism have been found to exacerbate common symptoms associated with autism, such as sleep problems and sensory sensitivities, having effective strategies to manage anxiety and stress may be particularly beneficial for autistic individuals. Mindfulness-based therapies have been increasingly recognized as promising interventions to reduce stress and anxiety, and improve mental health in individuals with and without autism. Several studies of individuals without autism have demonstrated that remote digital mindfulness training is equally as effective as traditional in-person mindfulness training in reducing stress and anxiety and enhancing well-being. However, there is little research investigating remote app-based mindfulness training for autistic individuals, which could be especially beneficial with this population due to anxiety and other constraints that make in-person training less feasible.

The primary objective is to assess efficacy of a six-week remote self-guided mindfulness intervention in reducing anxiety and stress in autistic adults. Autistic adults were invited to participate in a remote app-based mindfulness study where participants use their smartphones to complete the six-week structured mindfulness intervention. Participants were block randomized (based on initial trait anxiety scores) to either an intervention group or a wait-list control group. The intervention group immediately received the online mindfulness intervention. The wait-list control group received the same intervention program six-weeks later. All sessions and assessments were delivered online; thus participants were allowed maximal flexibility in participating in this fully remote intervention.

Self-reported levels of stress, anxiety, positive and negative emotions, and trait/dispositional mindfulness were measured at four time-points throughout the study: before the intervention, half-way through (at 3 weeks), after the intervention, and at follow-up (6 weeks after the end of the intervention). The wait-list control group was assessed at two additional time-points: before they began their waiting period and half-way through their waiting period (at 3 weeks). The primary aim of the study is to compare between-group (and secondarily, within-group) outcome measures to determine whether stress and anxiety levels decrease after the mindfulness intervention and whether they decrease above and beyond any decreases experienced by the wait-list control group.

Additionally, the study aims to:

* Determine whether and how changes in mindfulness are associated with changes in anxiety and stress, over the course of the intervention, including whether there is a negative association of mindfulness with stress and anxiety. In using two different measures of mindfulness the specific components of mindfulness can be examined that appear to be most likely to change and most likely to be (negatively) associated with stress and anxiety.
* Assess the feasibility of such a remote intervention with this sample of autistic adults by examining:

  * percentages of individuals in each group (intervention and wait-list control) who complete various stages of the intervention (e.g., post-test surveys, follow-up surveys).
  * percentages of individuals in each group (intervention and wait-list control) who complete all of the intervention activities, as well as those who complete at least a certain percentage (e.g. 50% and 75%) of the intervention activities.
* Examine who seems to benefit most from the intervention (by demographic variables, autistic traits, and other baseline measures obtained).

The aim is to have approximately 30 participants per group participate in the intervention and complete follow-up surveys. Individuals initially completed screening questionnaires to determine study eligibility. Eligible individuals were then given baseline measures, which included the outcome measures as well as autistic characterization measures. Participants were then randomly assigned (through block randomization based on baseline trait anxiety scores) to either the intervention group or the wait-list control group.

After completing their pre-intervention surveys participants were instructed to download the Healthy Minds customized application for this study and were then given a start date for the six-week self-guided intervention. They received automated emails instructing them to complete the outcome measures at the time-points specified above.

The intervention consisted of a customized version of the Healthy Minds app, with six-weeks of alternating didactic 'lessons' (each up to 7 minutes in length) and mindfulness 'practices' (either 10 minutes or 15 minutes in length- as chosen by the participant). There were a total of 29 lessons and practices that were part of the structured curriculum. Other optional practices were included on the app as well. Participants were instructed to listen to (at least) one activity per day for 5 days per week, for 6 weeks. They were told that it was suggested (but not required) that they listen to the activities in order, that they could re-listen to activities as they desired, and that they could listen to the optional practices as they saw fit.

Findings from this intervention will provide important information about the feasibility of remote app-based mindfulness training for autistic adults and the potential of remote app-based mindfulness training to reduce stress and anxiety in this population.

ELIGIBILITY:
Inclusion Criteria:

* Daily access to smartphone
* Professional diagnosis of autism spectrum disorder

Exclusion Criteria:

* Non-corrected hearing impairment (if it impacts their ability to listen to the app)
* Far below average nonverbal intellectual ability: 2 standard deviations below the mean on the Test My Brain, matrix reasoning subtest (a validated and normed proxy for nonverbal IQ)
* Listening comprehension skills that may compromise one's ability to understand the lessons and practices in the app: Below 60% correct on the Listening Comprehension measure (created for this study, based on language used in the Healthy Minds app)
* Ever taken part in a meditation retreat
* Engaged in meditation practice at least once per week over the past year
* Used Healthy Minds app ever
* Prior training with a meditation teacher (other than an introductory course)
* Practiced meditation daily for the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory for Adults | 6 Weeks
  40-item self-report assessing both state anxiety (20 items) and trait anxiety (20 items) on a 4-point Likert scale. Total trait anxiety scores range from 20 to 80. Total state anxiety scores range from 20 to 80. Higher scores are indicative of a greater level of anxiety.
Patient-Reported Outcomes Measurement Information System [PROMIS] Anxiety Short Form | 6 weeks
  8-item self-report measure of anxiety, on a 5-point Likert scale. Raw scores range from 8 to 40, with higher scores indicating more anxiety.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory for Adults | 12 Weeks
  40-item self-report assessing both state anxiety (20 items) and trait anxiety (20 items) on a 4-point Likert scale. Total trait anxiety scores range from 20 to 80. Total state anxiety scores range from 20 to 80. Higher scores are indicative of a greater level of anxiety.
Patient-Reported Outcomes Measurement Information System [PROMIS] Anxiety Short Form | 12 weeks
  8-item self-report measure of anxiety, on a 5-point Likert scale. Raw scores range from 8 to 40, with higher scores indicating more anxiety.
Perceived Stress Scale | 6 weeks
  10-item self-report measure of stress, on a 5-point Likert scale. Scores range from 0 to 40. Higher scores signify more stress.
Perceived Stress Scale | 12 weeks
  10-item self-report measure of stress, on a 5-point Likert scale. Scores range from 0 to 40. Higher scores signify more stress.
Positive and Negative Affect Schedule, Short Form | 6 weeks
  20-item self-report of 10 positive and 10 negative emotions, on a 5-point Likert scale, resulting in both a positive and a negative affect score. Scores for each scale range from 10-50, with higher scores on the Positive Affect Score indicating a greater degree of positive emotions, and higher scores on the Negative Affect Score indicating a greater degree of negative emotions.
Positive and Negative Affect Schedule, Short Form | 12 weeks
  20-item self-report of 10 positive and 10 negative emotions, on a 5-point Likert scale, resulting in both a positive and a negative affect score. Scores for each scale range from 10-50, with higher scores on the Positive Affect Score indicating a greater degree of positive emotions, and higher scores on the Negative Affect Score indicating a greater degree of negative emotions.

OTHER OUTCOMES:
Mindfulness Attention Awareness Scale | 3 weeks
  15-item self-report assessing trait mindfulness, on a 6-point Likert scale. Raw scores range from 15 to 90, with higher scores indicating more mindfulness.
Mindfulness Attention Awareness Scale | 6 weeks
  15-item self-report assessing trait mindfulness, on a 6-point Likert scale. Raw scores range from 15 to 90, with higher scores indicating more mindfulness.
Mindfulness Attention Awareness Scale | 12 weeks
  15-item self-report assessing trait mindfulness, on a 6-point Likert scale. Raw scores range from 15 to 90, with higher scores indicating more mindfulness.
Five Factor Mindfulness Questionnaire -Short Form | 3 weeks
  15-item self-report measure of 5 aspects of trait mindfulness, using a 5-point Likert scale. The total raw score ranges from 15 to 75. The raw scores of each of the 5 subscales range from 3 to 15. Higher scores indicate greater levels of trait mindfulness.
Five Factor Mindfulness Questionnaire -Short Form | 6 weeks
  15-item self-report measure of 5 aspects of trait mindfulness, using a 5-point Likert scale. The total raw score ranges from 15 to 75. The raw scores of each of the 5 subscales range from 3 to 15. Higher scores indicate greater levels of trait mindfulness.
Five Factor Mindfulness Questionnaire -Short Form | 12 weeks
  15-item self-report measure of 5 aspects of trait mindfulness, using a 5-point Likert scale. The total raw score ranges from 15 to 75. The raw scores of each of the 5 subscales range from 3 to 15. Higher scores indicate greater levels of trait mindfulness.
State-Trait Anxiety Inventory for Adults | 3 Weeks
  40-item self-report assessing both state anxiety (20 items) and trait anxiety (20 items) on a 4-point Likert scale. Total trait anxiety scores range from 20 to 80. Total state anxiety scores range from 20 to 80. Higher scores are indicative of a greater level of anxiety.
Patient-Reported Outcomes Measurement Information System [PROMIS] Anxiety Short Form | 3 weeks
  8-item self-report measure of anxiety, on a 5-point Likert scale. Raw scores range from 8 to 40, with higher scores indicating more anxiety.
Perceived Stress Scale | 3 weeks
  10-item self-report measure of stress, on a 5-point Likert scale. Scores range from 0 to 40. Higher scores signify more stress.
Positive and Negative Affect Schedule, Short Form | 3 weeks
  20-item self-report of 10 positive and 10 negative emotions, on a 5-point Likert scale, resulting in both a positive and a negative affect score. Scores for each scale range from 10-50, with higher scores on the Positive Affect Score indicating a greater degree of positive emotions, and higher scores on the Negative Affect Score indicating a greater degree of negative emotions.

CONTACTS AND LOCATIONS:
Overall Officials: John DE Gabrieli, PhD, Principal Investigator — Massachusetts Institute of Technology; Liron Rozenkrantz, PhD, Study Director — Massachusetts Institute of Technology
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to results in a publication will be available upon request to approved researchers.
Supporting Information: Study Protocol
Time Frame: De-identified data will be available upon request starting 6 months after publication and will remain available for 3 years.
Access Criteria: Data requests should be submitted to Cindy Li at cindyeli@mit.edu including a description of study aims as well as how the data will be utilized. Requests will be reviewed by the team and secure access to the requested data will be provided in the form of downloadable materials.